CLINICAL TRIAL: NCT05697575
Title: Non-interventional Observational Study to Evaluate the Efficacy and Safety of Non-immune Staphylokinase in Reperfusion Therapy of Ischemic Stroke in Routine Clinical Practice
Brief Title: Non-immunogenic Staphylokinase in Reperfusion Therapy of Ischemic Stroke in Routine Clinical Practice
Acronym: REPIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Society for Neurosonology and Cerebral Circulation (Other)
Responsible Party: Sponsor
Other Study IDs: REPIN-Forte
Record Dates: First submitted 2023-01-14; First posted 2023-01-26 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Acute Stroke
Keywords: stroke thrombolysis; acute ischemic stroke; reperfusion
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will collect data from aged 18 to 85 years with a diagnosis of acute stroke, who received thrombolytic treatment with a new agent, nonimmunogenic staphylokinase. Outcomes will be checked for safety and compared to the results of treatment with the other thrombolytic drug, alteplase.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 ;
* Diagnosis of acute ischemic stroke eligible for thrombolytic therapy;
* Thrombolytic therapy with the drug "non-immunogenic staphylokinase" is planned or has already been performed.

Exclusion Criteria:

* Individual intolerance or known hypersensitivity to a recombinant protein containing the amino acid sequence of staphylokinase;
* The presence of a contraindication to thrombolytic therapy of ischemic stroke;
* Pregnancy or lactation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 18 to 85 years (inclusive), who meet the inclusion criteria and do not have contraindications for thrombolysis, with a diagnosis of acute ischemic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of intracerebral hemorrhage | 36 hours
  Number and proportion of intracerebral bleeding of any type, which occurs as a complication of thrombolytic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Igor A Voznjuk, Prof, Study Director — First St. Petersburg State Medical University named after I.P. Pavlov
Locations (1):
- St. Petersburg Research Institute of Emergency Medicine named after I.I. Janelidze, Saint Petersburg, Russia